CLINICAL TRIAL: NCT03994003
Title: BIOmarkers and PREDISC Diagnostic Evaluation for Patients With Suspected Transient Ischemic Attacks: the BIOPREDISC- TIA SWISS Cohort Study
Brief Title: BIO-PREDISC-TIA SWISS Cohort Study
Acronym: PREDISC
Status: Completed | Type: Observational
Sponsor: Dr. med. Carlo Cereda (Other Government)
Collaborators: Ente Ospedaliero Cantonale, Bellinzona (Other)
Responsible Party: Sponsor-Investigator, Dr. med. Carlo Cereda, MD Capo Servizio, Ospedale Civico, Lugano
Organization: Ospedale Civico, Lugano (Other Government)
Other Study IDs: EOC.NSISU.4.12.99
Record Dates: First submitted 2019-06-19; First posted 2019-06-21 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Cerebrovascular Disease, Ischemic Stroke
MeSH Terms: conditions — Cerebrovascular Disorders; Ischemic Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — MiRNA will be isolated from whole blood collected in PAXgene tubes (BD/PreAnalytiX, Franklin Lakes, NJ). PAXgene tubes contain an RNA stabilizing reagent that acts at time of blood draw to prevent RNA degradation. RNA in whole blood is derived mainly from peripheral blood cells (monocytes, neutrophils, T cells, B cells, and megakaryocytes).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This research project aims at contributing to improve TIA diagnosis and management by using PREDISC scores and specific biomarkers thought to have elevated levels in TIA patients. A swift and accurate TIA diagnosis allows starting treatment of the patient adequately and shortly after the event. The shorter the time between the event and treatment onset, the better the outcome. This approach will be an important step forward in TIA diagnosis and management, similarly to acute coronary syndrome as discussed above.

ELIGIBILITY:
Inclusion Criteria:

* Patients with suspected TIA (defined as the acute onset of focal neurological symptoms lasting <24 h and presumed to be caused by brain ischemia at the time of referral) within 48 h of symptoms onset.

  * At least 18 years old.
  * Having given their Informed Consent.

Exclusion Criteria:

* · Patients with ocular TIA (Amaurosis fugax).

  * Patients that still have neurological deficits at the moment of inclusion.
  * Contraindication to perform MRI.
  * For women: pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with suspected TIA (defined as the acute onset of focal neurological symptoms lasting <24 h and presumed to be caused by brain ischemia at the time of referral) within 48 h of symptoms onset.
Sampling Method: Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2017-08-04 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Levels of specific biomarkers (Platelet Basic Protein (PBP), ceruloplasmin, microRNAs, exosomal particles) in patients with suspected TIA. | 1 year
  Diagnostic performance according to PREDISC scale

CONTACTS AND LOCATIONS:
Overall Officials: Carlo Cereda, MD, Study Director — Neurocentro della Svizzera Italiana Ospedale Regionale di Lugano
Locations (2):
- Switzerland (2):
  - Centre hospitalier Vaudois, Lausanne, Canton of Vaud
  - Ospedale Regionale di Lugano, Lugano, Canton Ticino